CLINICAL TRIAL: NCT03066505
Title: A Randomized, Double-blind, Sham-controlled Pilot Study to Evaluate the Treatment Efficacy of Magnetic EEG/ECG-Guided Resonance Therapy (MeRT) in College Students With Attention Deficit Hyperactivity Disorder.
Brief Title: A Randomized, Double-blind, Sham-controlled Pilot Study to Evaluate the Treatment Efficacy of Magnetic EEG/ECG-Guided Resonance Therapy (MeRT) in College Students With ADHD
Acronym: MeRT-USC-009
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wave Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MeRT-USC-009
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Sixteen (16) subjects will receive active treatment with MeRT and the other 15 with sham. Subjects in each study group will be treated 30 min a day, 5 days a week for 4 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects and clinicians will be blind to treatment condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active MeRT Treatment (Active Comparator): Active treatment will consist of 6 seconds a minute for 30 minutes a day, 5 days a week for 4 weeks.
  Interventions: Device: Active MeRT Treatment
- Sham MeRT Treatment (Sham Comparator): Sham treatment will consist of 6 seconds a minute for 30 minutes a day, 5 days a week for 4 weeks. Sham treatment mimicks same noise and sensation of active treatment but provides no treatment.
  Interventions: Device: Sham MeRT Treatment

INTERVENTIONS:
Device: Active MeRT Treatment — A personalized biometrics-guided protocol known as magnetic EEG/EKG resonance therapy (MeRT) treatment that is tailored specifically to each patient's higher harmonic frequency of heart rate, which is nearest to the characteristic frequency of alpha EEG frequency.
  Other Names: rTMS Active Stimulator
  Arms: Active MeRT Treatment
Device: Sham MeRT Treatment — A personalized biometrics-guided protocol similar to MeRT treatment that mimics magnetic EEG/EKG resonance therapy (MeRT) but does not emit active stimulation.
  Other Names: rTMS Sham Stimulator
  Arms: Sham MeRT Treatment

SUMMARY:
This pilot study is a randomized, double-blind, sham-controlled study designed to evaluate the efficacy of Magnetic EEG/ECG-Guided Resonance Therapy (MeRT) in college students with ADHD. A total of 40 subjects will be treated.

DETAILED DESCRIPTION:
This pilot study is a randomized, double-blind, sham-controlled study designed to evaluate the efficacy of Magnetic EEG/ECG-Guided Resonance Therapy (MeRT) in college students with ADHD. A total of 40 subjects will be treated.

Twenty (20) subjects will receive active treatment with MeRT and the other 20 with sham. Subjects in each study group will be treated 30 min a day, 5 days a week for 4 weeks. This is known as Phase 1. During this study period, subjects and clinicians will be blind to treatment condition.

Subjects will be recruited from a flyer describing the study. The flyer will be posted at the Kortschak Center for Learning and Creativity, the McKay Center, and through Student Counseling Services in the Engemann Student Health Center. In addition, students who have been diagnosed with ADHD and have been seen at one of these facilities for ADHD may be provided contact information for the study.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to qualify for enrollment into the study:

1. College student 18-25 years of age
2. Diagnosed with ADHD using the standardized clinical interview and supported by the Pearson Quotient ADHD System and Conners Adult ADHD Rating Scales (CAARS)
3. Willing and able to adhere to the treatment schedule and all required study visits

Exclusion Criteria:

Subjects will be excluded from study participation if one of the following exclusion criteria applies:

1. Pregnant or trying to become pregnant; negative urine pregnancy test at screening will be required of females of child-bearing potential
2. Any antipsychotic or anticonvulsant medication.
3. Any type of rTMS treatment within 3 months prior to the screening visit
4. Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, stents, or electrodes) or any other metal object within or near the head, excluding the mouth, which cannot be safely removed
5. Any condition which in the judgment of the investigator would prevent the subject from completing the study
6. Any seizure history within the past 10 years
7. EEG abnormalities including indications of risk of seizure, i.e., abnormal focal or general slowing in spikes during the EEG recording
8. Unstable medical conditions such as uncontrolled endocrine, hepatic, cardiac, pulmonary and/or renal disorders.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

PRIMARY OUTCOMES:
Pearson Quotient ADHD System | Four weeks.
  Changes in Pearson Quotient ADHD System; arithmetic changes in Pearson Quotient ADHD System score between time points at baseline and end of week 4.
Conners Adult ADHD Rating Scales (CAARS) | Four weeks.
  Changes in Conners Adult ADHD Rating Scales (CAARS) ; arithmetic changes in Conners Adult ADHD Rating Scales (CAARS) total score between time points at baseline and end of week 4.
Electroencephalogram (EEG) Assessment | Four weeks.
  Changes in electroencephalogram (EEG) will be assessed at baseline, week 2 and end of week 4.

SECONDARY OUTCOMES:
Rivermead Post Concussion Symptoms Questionnaire (RPQ) | Four weeks.
  Changes in Rivermead Post Concussion Symptoms Questionnaire (RPQ); arithmetic changes in Rivermead Post-Concussion Symptoms Questionnaire (RPQ-16) total score between time points at baseline and end of week 4.

OTHER OUTCOMES:
Safety Outcomes assessed by Arithmetic number of Adverse Events (AEs) and Serious Adverse Events (SAEs). | Four weeks.
  Arithmetic number of Adverse Events (AEs) and Serious Adverse Events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Charles Liu, MD, PhD, Principal Investigator — University of Southern California Neurorestoration Center
Locations (1):
- USC Neurorestoration Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No